CLINICAL TRIAL: NCT04889456
Title: Implementation of Optimized and Standardized Surgical Technique for Right Sided Colon Cancer: a Prospective Interventional Sequential Cohort Study With a Transition Period
Brief Title: Standardizing Right Hemicolectomy for Colon Cancer
Acronym: Right
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Prof. dr. P.J. Tanis, colorectal surgeon (Unknown); Dr. B.R. Toorenvliet, colorectal surgeon (Unknown); D. Miskovic, St Marks hospital London, UK (Unknown); S. Benz, Klinikverbund SuedWest, Böblingen, Germany (Unknown); F. Aigner, Krankenhaus der Barmherzigen Bruder, Graz, Austria (Unknown); C.A. Bertelsen, Hillerød University Hospital, Copenhagen, Denmark (Unknown); Drs. A.A.J. Grüter (Unknown); Dr. U.K. Coblijn (Unknown); Dr. H.L. van Westreenen (Unknown); Dr. C. Sietses (Unknown); Prof. dr. E.C.J. Consten (Unknown); Dr. A.W.H. van de Ven (Unknown); Dr. P. van Duijvendijk (Unknown); Dr. S. van Aalten (Unknown); Dr. F. den Boer (Unknown); Dr. J.W.A. Leijtens (Unknown); Dr. C. Hoff (Unknown); Dr. O. van Ruler (Unknown); Dr. G. D. Slooter (Unknown); Prof. dr. J. Lange (Unknown); Prof. dr. G.J. Kleinrensink (Unknown)
Responsible Party: Principal Investigator, Jurriaan B. Tuynman, Dr, Amsterdam UMC, location VUmc
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021.0273
Record Dates: First submitted 2021-04-30; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Colonic Carcinoma; Laparoscopic Right Hemicolectomy; Standardisation; Training; Delphi Study; Implementation; Consolidation; Assessment
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective interventional sequential cohort study with a transition period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surgical variations laparoscopic right hemicolectomy (No Intervention)
- Implementing standardised laparoscopic right hemicolectomy with proctoring (Active Comparator)
  Interventions: Procedure: Implementation standardised laparoscopic right hemicolectomy with proctoring
- Implementing standardised laparoscopic right hemicolectomy without proctoring (Active Comparator)
  Interventions: Procedure: Implementation standardised laparoscopic right hemicolectomy without proctoring

INTERVENTIONS:
Procedure: Implementation standardised laparoscopic right hemicolectomy with proctoring — Implementation standardised laparoscopic right hemicolectomy with proctoring
  Arms: Implementing standardised laparoscopic right hemicolectomy with proctoring
Procedure: Implementation standardised laparoscopic right hemicolectomy without proctoring — Implementation standardised laparoscopic right hemicolectomy without proctoring
  Arms: Implementing standardised laparoscopic right hemicolectomy without proctoring

SUMMARY:
A surgical intervention might be highly variable amongst surgeons and centers. This variability has a potential relevance concerning clinical outcomes.

For right-sided colon cancer, the laparoscopic right hemicolectomy (LRHC) knows substantial variation. Especially since the surgical technique has been evolving during the latest decade with the introduction of intracorporeal anastomosis, a dissection technique within the correct embryological planes (complete mesocolic excision) and central vascular ligation of the segmental branches at its origin, resulting in an optimal lymph node dissection.

Given the insights from recent studies showing the association between quality of surgery and relevant clinical outcomes, there is a great need for a formative quality assessment of LRHC. Detailed objective assessment of the LRHC is currently not performed in clinical practice nor in surgical training. Quality assessment of LRHC has great potential to improve surgical training and furthermore, implementation of a standardized technique will ultimately lead to better quality of care for patients suffering from right-sided colon cancer.

The main objective of this study is to improve surgical outcomes for patient with right-sided colon cancer by a prospective sequential interventional cohort study that aims to standardize the surgical technique with subsequent controlled implementation after standardized review of the current practice in a nationwide multicenter setting. The primary endpoint is the 30-day morbidity according to the Clavien-Dindo classification system.

DETAILED DESCRIPTION:
1. Prospective mapping of current practice with surgical variations in laparoscopic right hemicolectomy (total duration of inclusion 3 months) N= 40 centers N = 310 videos

   1. METC approval for the use of anonymized videos of a laparoscopic procedure and collection of corresponding clinical outcomes.
   2. Approaching hospitals for participation (high volume centers (50+ colon cancers).
   3. Prospective inclusion of consecutive patients undergoing laparoscopic right hemicolectomy in the participating hospitals in three months.
2. Development of Standard Laparoscopic Right Hemicolectomy: an (inter)national Delphi study

   1. Approaching specialists to participate in the Delphi method (from participating hospitals in step 1).
   2. Identification of crucial steps and measures according to literature and expert's opinion (Delphi method).
   3. Documentation of steps and the order in which they need to be performed, development of a competency assessment tool (CAT).
3. Skills center training facility

   a. Training the participating surgeons in the method of the standardized laparoscopic right hemicolectomy, as consented in the Delphi method.
4. Implementation of the standardized laparoscopic right hemicolectomy with proctoring during another period with prospective inclusion of consecutive patients with collection of surgical videos in all participating hospitals (N=40 centers, total 310 videos)

   1. Rating videos.
   2. Comparing with pre-implementation performance based on outcome measures reflecting oncological quality of surgery, and 30-day clinical outcomes.
   3. Comparing with pre-implementation performance based on the long-term outcomes. (3-year DFS and 5-year OS).
5. Implementing standardised lap right hemicolectomy (after learning curve without proctoring)

   1. Consecutive inclusion of patients (n=310)
   2. CT imaging
   3. Video analysis
   4. Competency analysis
   5. Variation analysis
   6. Clinico pathological data

ELIGIBILITY:
Inclusion Criteria:

* Planned laparoscopic (extended) right hemicolectomy for colon cancer of the caecum, ascending colon or hepatic flexure;
* Age above 18 years;
* cTNM stage 1-3 (CT-staged);
* No prior midline or transverse laparotomy;
* ASA1-3;
* No immune modulating medication.

Exclusion Criteria:

* cT4b;
* Perforated disease;
* Acute obstruction;
* Emergency operation;
* Appendiceal cancer;
* Other primary malignancy treated within 5 years from diagnosis of colon cancer, except for curatively treated prostate, breast, skin and cervical cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 930 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
30-day morbidity with Clavien-Dindo grading | 30 days

SECONDARY OUTCOMES:
Intraoperative complications (i.e. vascular injury) | 1 day
Conversion rate from laparoscopic to open surgery | 1 day
Operative time | 1 day
Blood loss | 1 day
Validated assessment of plane of dissection | 1 day
  Assessment according to a competency assessment tool (CAT) for laparoscopic right hemicolectomy. This tool will be created during phase 2 using the Delphi method.
Validated assessment of level of vascular ligation | 1 day
  Assessment according to a competency assessment tool (CAT) for laparoscopic right hemicolectomy. This tool will be created during phase 2 using the Delphi method.
Grading of the resection specimen according to Benz et al. 2019 | 1 day
Total lymph node count | 1 day
Number of resected positive lymph nodes | 1 day
Resection margins | 1 day
  Radicality of resection margin of the specimen, as assessed by the pathologist.
Completeness of mesocolic excision based on postoperative CT imaging | 1 day
Locoregional recurrence | 3 years
Distant metastasis | 3 years
3-year disease free survival (DFS) | 3 years
5-year overall survival (OS) | 5 years
Long term morbidity: incisional hernia, adhesion related small bowel obstruction, readmissions, reinterventions | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gruter AAJ, Coblijn UK, Toorenvliet BR, Tanis PJ, Tuynman JB; Right Collaborators Group. National implementation of an optimal standardised technique for right-sided colon cancer: protocol of an interventional sequential cohort study (Right study). Tech Coloproctol. 2023 Nov;27(11):1083-1090. doi: 10.1007/s10151-023-02801-6. Epub 2023 Apr 25. PMID 37097330